CLINICAL TRIAL: NCT05352230
Title: Continuous Glucose Monitoring (CGM) in Kidney-Transplanted Adults
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: cessation of funds for study activities
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Orlando M. Gutierrez, MD, MMSc, Professor of Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-300009227
Record Dates: First submitted 2022-04-20; First posted 2022-04-28 (Actual); Results first posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus; Kidney Transplant; Complications
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Continue Glucose Monitoring (CGM) (Active Comparator): External diabetes device glucose sensor that measures interstitial glucose levels every minute
  Interventions: Device: Free style libre-2
- Glucometer (Other): Device that measures capillary blood glucose levels
  Interventions: Device: Free style libre-2

INTERVENTIONS:
Device: Free style libre-2 — A cross-over design will allow estimation of feasibility and acceptability of patients using CGM vs patients using blood glucose meter monitoring (conventional therapy). The study will consist on two phases, the first will last three months, then it will be a two months of washout period followed by the crossover, then the second phase will last another three months. Patients in the conventional therapy group will also use masked CGM (CGM professional) during the first two and last two weeks of their study phase with the purpose of collecting CGM-parameters information. The cross over randomization will be stratified by donor type (live vs deceased) using a web-based randomization tool. During the washout period the patients will continue using blood glucose meter monitoring

SUMMARY:
Pre-existing diabetes prior KT and Early Post-Transplant Hyperglycemia (PTRH) defined as a fasting blood glucose greater than or equal to 126 mg/dL or random glucose greater than or equal to 200 mg/dL or requirement of insulin during the first 45 days after KT has been associated with increased risks of post-transplant organ rejection. PTRH has also been associated to high infection rates, and in some cases, early mortality. The use of continuous glucose monitoring (CGM) compared with blood glucose meter monitoring in non-transplant patients with diabetes resulted in lower HbA1C by 0.4 to 0.5% within the first three months of use without major changes in patients' antidiabetic regimen, possibly due to patients become more conscious about their diabetes status and diet. CGM free style libre-2 measures the interstitial fluid every minute and their glucose sensors are replaced every two weeks. To our knowledge there are no studies that assess the role of CGM in improving glycemic and transplant outcomes in solid organ transplant patients, mainly because access to CGM is often limited by inadequate health insurance coverage or high out-of-pocket costs.

The investigators hypothesize that the intervention will be feasible and acceptable to patients, and our overarching hypothesis is that patients who wear a CGM will have better glycemic control, using a proxy measure of lower fructosamine/albumin ratio and better CGM-parameters, compared to those who did not wear it. Fructosamine represents the average glycemia for the 2 to 3 weeks prior. It is useful in any situation where glycemic control needs to be assessed over a period shorter than a month and in cases involving interference in the HbA1C measurement such as in adults with KT due to shorter red blood cell lifespan related to anemia of chronic disease. Fructosamine values vary in relation to the serum albumin concentration, which makes the fructosamine/albumin ratio the ideal physiologic measure for this pilot study . The investigators also hypothesize that patients who wear a CGM will have less microalbuminuria compared to those who did not wear it.

DETAILED DESCRIPTION:
Diabetes is a leading cause of end-stage renal disease, which is treated by undergoing kidney transplantation. Glycemic control post-transplantation is complicated for the diabetic population by a complicated medication regimen that suppresses immunologically-driven graft loss but increases glucose levels. Hyperglycemia in this transplant population results in transplant failure. Improving glycemic control in the diabetic kidney transplant population may decrease kidney transplantation failure rates. Continuous glucose monitors have been shown to improve glycemic control among insulin-dependent diabetics. Therefore, the investigators aim to assess the feasibility and acceptance of continuous glucose monitoring among diabetic kidney transplant patients.

This is an open-label, randomized, crossover design study comparing diabetic, kidney-transplant recipients managing their diabetes with a continuous glucose monitor or glucometer. Eligible participants will engage study staff during regularly scheduled, standard of care, post-operative visits. Utilization of the CGM will be assess to determine the feasibility of CGM usage in this population. Participants will complete validated quality-of-life surveys (Diabetes Treatment Satisfaction Questionnaire (DSTQ) and Hypoglycemic Confidence Scale (HSC)) throughout the 32 weeks study regimen to inform the acceptability of CGM usage. Glucose records, provided by glucose meters and CGMs that report glucose readings to either the participant or clinic will be leveraged to estimate if CGM usage decreases hyperglycemia among diabetic kidney-transplant recipients.

Results from this study will be foundational towards assessing if CGM usage improves glycemic control among diabetic kidney-transplant recipients, improves transplant outcomes and, hopefully, triggering health insurance providers to reassess the return on investment of subsidizing continuous glucose monitoring in the kidney-transplant population.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years
* patients with history of diabetes (either T1D, T2D or atypical diabetes forms)
* patients could be on insulin or not before transplantation

Exclusion Criteria:

* kidney-pancreas transplanted participants
* not currently using CGM (but could have used a year prior the transplant)
* mental conditions that prevent continuing with the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-05-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UAB Hospital, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of ten participants were screened for eligibilty between April of 2023 and October of 2023
Pre-assignment Details: A total of 4 participants were randomized. Of those not randomized, 6 did not meet inclusion/exclusion criteria
Groups:
- Continue Glucose Monitoring (CGM), Then Standard Glucometer: External diabetes device glucose sensor that measures interstitial glucose levels every minute
  Free style libre-2: A cross-over design will allow estimation of feasibility and acceptability of patients using CGM vs patients using blood glucose meter monitoring (conventional therapy). The study will consist on two phases, the first will last three months, then it will be a two months of washout period followed by the crossover, then the second phase will last another three months. Patients in the conventional therapy group will also use masked CGM (CGM professional) during the first two and last two weeks of their study phase with the purpose of collecting CGM-parameters information. The cross over randomization will be stratified by donor type (live vs deceased) using a web-based randomization tool. During the washout period the patients will continue using blood glucose meter monitoring
- Glucometer, Then Continuous Gluose Monitoring (CGM): Device that measures capillary blood glucose levels
  Free style libre-2: A cross-over design will allow estimation of feasibility and acceptability of patients using CGM vs patients using blood glucose meter monitoring (conventional therapy). The study will consist on two phases, the first will last three months, then it will be a two months of washout period followed by the crossover, then the second phase will last another three months. Patients in the conventional therapy group will also use masked CGM (CGM professional) during the first two and last two weeks of their study phase with the purpose of collecting CGM-parameters information. The cross over randomization will be stratified by donor type (live vs deceased) using a web-based randomization tool. During the washout period the patients will continue using blood glucose meter monitoring
Period: First Intervention (3 Months)
Arm/Group | Continue Glucose Monitoring (CGM), Then Standard Glucometer | Glucometer, Then Continuous Gluose Monitoring (CGM)
Started | 2 | 2
Completed | 0 | 0
Not Completed | 2 | 2
Not completed — study terminated | 2 | 2
Period: Washout (2 Months)
Arm/Group | Continue Glucose Monitoring (CGM), Then Standard Glucometer | Glucometer, Then Continuous Gluose Monitoring (CGM)
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0
Period: Second Intervention (3 Months)
Arm/Group | Continue Glucose Monitoring (CGM), Then Standard Glucometer | Glucometer, Then Continuous Gluose Monitoring (CGM)
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Continue Glucose Monitoring (CGM), Then Glucometer: External diabetes device glucose sensor that measures interstitial glucose levels every minute for 12 weeks, followed by standard glucometer that measures capillary blood glucose levels for 12 weeks with an 8 week wash out period in between
- Glucometer, Then Continuous Glucose Monitoring (CGM): Device that measures capillary blood glucose levels for 12 weeks followed by an external diabetes device glucose sensor that measures interstitial glucose levels every minute for 12 weeks with an 8 week wash out period in between
- Total: Total of all reporting groups
Arm/Group | Continue Glucose Monitoring (CGM), Then Glucometer | Glucometer, Then Continuous Glucose Monitoring (CGM) | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (1) | 58 (4) | 55 (3)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex
  Participants
    Female | 1 | 1 | 2
    Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — race
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 2 | 2 | 4
    White | 0 | 0 | 0
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Compliance
Description: To determine the feasibility and acceptance of CGM in adults with diabetes who underwent kidney transplantation compared to those who use glucometers.
Time Frame: 32 weeks
Population: Data were not collected due to study termination prior to participants' assessment at the pre-specified time points
Groups:
- Continue Glucose Monitoring (CGM), Then Glucometer; Glucometer, Then Continuous Glucose Monitoring: External diabetes device glucose sensor that measures interstitial glucose levels every minute
  Free style libre-2: A cross-over design will allow estimation of feasibility and acceptability of patients using CGM vs patients using blood glucose meter monitoring (conventional therapy). The study will consist on two phases, the first will last three months, then it will be a two months of washout period followed by the crossover, then the second phase will last another three months. Patients in the conventional therapy group will also use masked CGM (CGM professional) during the first two and last two weeks of their study phase with the purpose of collecting CGM-parameters information. The cross over randomization will be stratified by donor type (live vs deceased) using a web-based randomization tool. During the washout period the patients will continue using blood glucose meter monitoring
Arm/Group | Continue Glucose Monitoring (CGM), Then Glucometer | Glucometer, Then Continuous Glucose Monitoring
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Fructosamine/Albumin Ratio
Description: glycemic marker
Time Frame: 20 weeks
Population: Data were not collected due to study termination prior to participants' assessment at the pre-specified time points
Groups:
- Glucometer, Then Continuous Glucose Monitoring: Device that measures capillary blood glucose levels
  Free style libre-2: A cross-over design will allow estimation of feasibility and acceptability of patients using CGM vs patients using blood glucose meter monitoring (conventional therapy). The study will consist on two phases, the first will last three months, then it will be a two months of washout period followed by the crossover, then the second phase will last another three months. Patients in the conventional therapy group will also use masked CGM (CGM professional) during the first two and last two weeks of their study phase with the purpose of collecting CGM-parameters information. The cross over randomization will be stratified by donor type (live vs deceased) using a web-based randomization tool. During the washout period the patients will continue using blood glucose meter monitoring
Arm/Group | Continue Glucose Monitoring (CGM), Then Glucometer | Glucometer, Then Continuous Glucose Monitoring
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Fructosamine/Albumin Ratio
Description: glycemic marker
Time Frame: 32 weeks
Population: Data were not collected due to study termination prior to participants' assessment at the pre-specified time points
Arm/Group | Continue Glucose Monitoring (CGM), Then Glucometer | Glucometer, Then Continuous Glucose Monitoring
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Microalbuminuria
Description: kidney function marker
Time Frame: 20 weeks
Population: study terminated early before outcomes are collected
Arm/Group | Continue Glucose Monitoring (CGM), Then Glucometer | Glucometer, Then Continuous Glucose Monitoring
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Microalbuminuria
Description: kidney function marker
Time Frame: 32 weeks
Population: Data were not collected due to study termination prior to participants' assessment at the pre-specified time points
Arm/Group | Continue Glucose Monitoring (CGM), Then Glucometer | Glucometer, Then Continuous Glucose Monitoring
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Glucose Management Indicator (GMI)
Description: glycemic marker
Time Frame: 20 weeks
Population: Data were not collected due to study termination prior to participants' assessment at the pre-specified time points
Arm/Group | Continue Glucose Monitoring (CGM), Then Glucometer | Glucometer, Then Continuous Glucose Monitoring
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Glucose Management Indicator (GMI)
Description: glycemic marker
Time Frame: 32 weeks
Population: Data were not collected due to study termination prior to participants' assessment at the pre-specified time points
Arm/Group | Continue Glucose Monitoring (CGM), Then Glucometer | Glucometer, Then Continuous Glucose Monitoring
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Time in Range (TIR) of 70 to 180 mg/dL
Description: glycemic marker
Time Frame: 20 weeks
Population: Data were not collected due to study termination prior to participants' assessment at the pre-specified time points
Arm/Group | Continue Glucose Monitoring (CGM), Then Glucometer | Glucometer, Then Continuous Glucose Monitoring
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Time in Range (TIR) of 70 to 180 mg/dL
Description: glycemic marker
Time Frame: 32 weeks
Population: Data were not collected due to study termination prior to participants' assessment at the pre-specified time points
Arm/Group | Continue Glucose Monitoring (CGM), Then Glucometer | Glucometer, Then Continuous Glucose Monitoring
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 33 weeks
Arm/Group | Continue Glucose Monitoring (CGM) | Glucometer
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-30): https://cdn.clinicaltrials.gov/large-docs/30/NCT05352230/Prot_SAP_002.pdf